CLINICAL TRIAL: NCT04556864
Title: Hemodynamic Impact on Critical Care Patients With Lung Damage Secondary to SARS-CoV-2 Infection
Brief Title: Hemodynamic Impact on Critical Care Patients With Lung Damage Secondary to COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Juan Victor Lorente (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor-Investigator, Juan Victor Lorente, Medical Doctor, Andalusian Network for Design and Translation of Advanced Therapies
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FAB-HEM-2020-01
Record Dates: First submitted 2020-09-12; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Hemodynamic Instability; ARDS, Human
Keywords: COVID; hemodynamic monitoring; ARDS
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Description Group: * For each patient included in the study, the secondary variables will be noted in the patient's data collection logbook.
  * This is followed by radial artery cannulation (if absent), and connection to the HemoSphere/EV1000 platform
  * After the daily visit, the PI/collaborating investigators (CI) will measure the clinical, treatment, and mechanical ventilation parameters of the patient during the last 24 hours.
  * Daily arterial analysis will be requested
  * This information collection process will be followed for 5 days. At the end of the information collection period, the IP will perform two downloads, the engineering download, and the standard download in which the values are monitored every 20 seconds.
  * These will be noted in the secondary variables of the data collection logbook, along with the patients' ICU discharge date.
  * In-hospital mortality will be monitored during admission to a conventional hospital ward.
  * Records will be closed upon discharge of the patient.

SUMMARY:
The aim of the present work is to describe the hemodynamic effects shown in patients with ARDS secondary to SARS-CoV-2 infection

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients that are classified as a "confirmed case" according to criteria established by the Spanish Ministry of Health in its Technical Document updated on March 31, 2020. This defines a "confirmed case" as a case that meets laboratory criteria (Positive PCR test for any of the SARS-CoV-2 genes).
* Patients admitted to ICU.
* Presence of Kirby index (PaFi) less than or equal to 300 mm Hg, with PEEP or CPAP greater than or equal to 5 cmH2O.
* Need for radial artery cannulation for hemodynamic monitoring and/or repeated monitoring of blood gases at the discretion of the responsible physician.
* Patients who agree (or a representative of the patient if sedated) to participate in study and who provide written informed consent.

Exclusion Criteria:

* Patients being treated with veno-venous or veno-arterial ECMO
* Patient with therapeutic restrictions due to life support
* Patient who presents a complication that requires surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS secondary to SARS-CoV-2 infection
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Total amount of hypotension | 5 days
  Hypotension will be defined as a hemodynamic event that occurs when the MAP falls below 65 mmHg for a minimum duration of 1 minute (3 consecutive recordings of 1 minute or more between two consecutive falls of the MAP).

SECONDARY OUTCOMES:
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor (Stroke volume) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor (Stroke volume variation) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor (Cardiac index) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor ( HPI) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor (Eadyn) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Minimally invasive hemodynamic monitoring and related variables obteined from HemoSphere platform with Acumen IQ sensor (dp/dt max,) | 5 days
  We will obtain hemodynamic data for the first 5 days after the patient enters the study
Presence of treatment with noradrenaline; presence of treatment with dobutamine, presence of treatment with other vasoactive/ionotropic/hypotensive drugs | 5 days
  start time, time of dose change, current dose
Furosemide treatment | Daily during 5 days
  dose/24 hours
Daily diuresis, daily water balance, accumulated water balance since ICU admission, daily parenteral nutrition volume, and daily enteral nutrition volume. | Daily during 5 days
  ml/24 h
Atrial fibrillation | 5 days
  Presence, start time and end time
Acute kidney injury | Daily during 5 days
  Presence and degree with KDIGO definition
Continuous renal replacement therapies | 5 days
  Start and end date/time, dialyzing flow, replacement flow, daily balance.
Need for Hemadsorption | 5 days
  Start and end date/time, blood flow.
Specific treatment for SARS-CoV2 (presence of tocilizumab, antimalarial drugs, antivirals) | 5 days
  Start and end date/time
Corticoid treatment. | 5 days
  Start and end date/time

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - 1. A.H. Juan Ramón Jiménez., Huelva, Andalusia
  - 5. Hospital Virgen de la Victoria, Málaga, Andalusia
  - 4. Hospital Universitario de Álava., Alava, Basque Country
  - 3. Hospital Universitario. Jerez de la Frontera., Jerez de la Frontera, Cádiz
  - 2. Hospital Universitario Infanta Leonor, Madrid